CLINICAL TRIAL: NCT03379597
Title: A 12-weeks Study to Evaluate the Dietary Fiber and Probiotics Treatment in Prevention and Intervention of Weight-gain and Cognitive Impairment of Schizophrenia or Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, Central South University, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WU201711BIO
Record Dates: First submitted 2017-11-29; First posted 2017-12-20 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: Schizophrenia; probiotics; cognitive impairment; Metabolic syndrome; clinical trail; Efficacy; Safety; Dietary fiber; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Cognitive Dysfunction; Metabolic Syndrome | interventions — Lacteol; Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Probiotics Group (Experimental): Probiotics add-on treatment :（live Combined Bifidobacterium, Lactobacillus and Enterococcus Capsules, Oral）, each capsule contain more then 1.0*10^7 CFU.
  Bifico: 840mg Bid.
  Interventions: Drug: Bifico (Live combined bifidobacterium,Lactobacillus and Enterococcus capsules, Oral)
- Control Group (No Intervention): No probiotics or dietary fiber group.
- Dietary fiber Group (Experimental): Prebiotics add-on treatment: dietary fibers compound powder, 30g bid
  Interventions: Dietary Supplement: Dietary fiber
- Dietary fiber Probiotics group (Experimental): Dietary fiber and probiotics group: receiving both Bifico 840mg Bid and dietary fiber 30g bid.
  Interventions: Drug: Bifico (Live combined bifidobacterium,Lactobacillus and Enterococcus capsules, Oral); Dietary Supplement: Dietary fiber

INTERVENTIONS:
Drug: Bifico (Live combined bifidobacterium,Lactobacillus and Enterococcus capsules, Oral) — Bifico 840mg Bid
  Arms: Dietary fiber Probiotics group; Probiotics Group
Dietary Supplement: Dietary fiber — dietary fiber compound powder 30g bid
  Arms: Dietary fiber Group; Dietary fiber Probiotics group

SUMMARY:
In this study, the investigators will evaluate the efficacy, safety and related mechanism of dietary fiber and probiotics alone and in combination as a add-on treatment in improving the antipsychotic induced weight gain, the cognitive impairment, and psychotic syndrome in schizophrenia or bipolar disorder patients. The study will recruit 100 schizophrenia or bipolar disorder patients who meet the criteria of DSM-5, and then randomized to 4 groups: probiotics group(PB group) dietary fiber group(FB group) probiotics plus dietary fiber group(PF group) and control group(CT group) for a 12-weeks clinical trail. The specific aims are to compare probiotics group versus controls on: 1) clinical core symptoms; 2) cognition;3)metabolic related markers.

DETAILED DESCRIPTION:
In this study, the investigators will evaluate the efficacy, safety and related mechanism of dietary fiber and probiotics alone and in combination as a add-on treatment in improving the antipsychotic induced weight gain, the cognitive impairment, and psychotic syndrome in schizophrenia or bipolar disorder patients. The study will recruit 100 schizophrenia or bipolar disorder patients who meet the criteria of DSM-5, and then randomized to 4 groups: probiotics group(PB group) dietary fiber group(FB group) probiotics plus dietary fiber group(PF group) and control group(CT group) for a 12-weeks clinical trail (20 patients per arm) for a 12-weeks clinical trail. Clinical efficacy and safety assessment will be done at screen/baseline, 4 week, 8 week and 12 week. The specific aims are to compare probiotics group versus controls on: 1) clinical core symptoms; 2) cognition; 3) metabolic related markers. Biological samples also will be collected, and stored to research related mechanisms. Clinical symptoms will be measured by the Positive and Negative Syndrome Scale,. Cognitive function will be assessed by the MATRICS Consensus Cognitive Battery.

The investigators hypothesize that: 1) dietary fiber and probiotics may improve cognitive impairment of patients with schizophrenia; 2) dietary fiber and probiotics could prevent the cognitive decline of patients with schizophrenia; 3)dietary fiber and probiotics may prevent the antipsychotics induced weight gain in patients with schizophrenia.4)dietary fiber and probiotics may alter oxidative stress indexes or inflammatory biomarkers thus influence the oxidative and inflammatory mechanism.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the Diagnostic and Statistical Manual (DSM-V) diagnostic criteria for schizophrenia or bipolar disorder;
2. Patients with a weight gain of more than 10% after taking antipsychotic medications;
3. Male and female with aged 18 to 65 years;
4. PANSS total score < 60 or HAMD-17 total score≤ 7 and YMRS total score<5;
5. Signed the study consent for participation;
6. Not allergy to probiotics or dietary fiber medicine
7. On stable medication and dosage for at least 3 months.

Exclusion Criteria:

1. Having history of substance dependence or abuse or whose symptoms are caused by the other diagnosable mental disorders;
2. Having history of traumatic brain injury, seizures or other known neurological or organic diseases of the central nervous system;
3. Taking antidepressants, stimulants, mood stabilizer or accepts electricity shock treatment;
4. Having current suicidal or homicidal thoughts or any safety concern by research staff that cannot be manage in an inpatient setting;
5. The routine blood tests showing abnormal renal, liver function;
6. Pregnant or lactating women.
7. No administration of any antibiotics in two mouths

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
MATRICS Consensus Cognitive Battery (MCCB) composite score | 12 weeks
  The investigators will use the MATRICS Consensus Cognitive Battery (MCCB) Composite score as primary cognitive outcome measure before and after treatment at different follow up point.
Body Mass Index | 12 weeks
  The body mass index (BMI) or Quetelet index is a value derived from the mass (weight) and height of an individual. The BMI is defined as the body mass divided by the square of the body height, and is universally expressed in units of kg/m2, resulting from mass in kilograms and height in metres.

SECONDARY OUTCOMES:
Positive And Negative Syndrome Scale (PANSS) | 12 weeks
  The change of Positive And Negative Syndrome Scale (PANSS) total, positive and negative symptoms before and after treatment at different follow up point.
Lipid metabolism related blood index | 12 weeks
  Other lipid metabolism related marker such as LDL,HDL,TG, CHO (all in mmol/L)
Physical exam index | 12 weeks
  Body weight related physical exam index: waist circumference,hip line (cm)
Hamilton Depression Scale and Young Manic Rating Scale (YMRS) | 12 weeks
  The change of total score of the Hamilton Depression Scale and the Young Manic Rating Scale (YMRS), used to measure mania and depression symptoms of bipolar disorder.

CONTACTS AND LOCATIONS:
Overall Officials: DongYu Kang, M.D., Principal Investigator — Central South University; SuJuan Li, M.D., Principal Investigator — Central South University; RenRong Wu, M.D. Ph.D., Principal Investigator — Central South University; Chenchen Liu, M.D., Principal Investigator — Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

REFERENCES:
- [Derived] Liu C, Kang D, Xiao J, Huang Y, Peng X, Wang W, Xie P, Yang Y, Zhao J, Wu R. Dietary fiber and probiotics for the treatment of atypical antipsychotic-induced metabolic side effects: study protocol for a randomized, double-blind, placebo-controlled trial. Trials. 2021 Feb 23;22(1):159. doi: 10.1186/s13063-021-05123-w. PMID 33622382